CLINICAL TRIAL: NCT07271069
Title: Real-world Effectiveness of Ozanimod in Patients With Steroid-Dependent Ulcerative Colitis: A Chart Review Study
Brief Title: Effectiveness of Ozanimod in Patients With Steroid-Dependent Ulcerative Colitis
Status: Not yet recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM047-1120
Record Dates: First submitted 2025-11-27; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ozanimod; Azathioprine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Group 1: Participants with ulcerative colitis receiving ozanimod
  Interventions: Drug: Ozanimod
- Group 2: Participants with ulcerative colitis receiving azathioprine
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Ozanimod — According to the product label
  Groups: Group 1
Drug: Azathioprine — According to the product label
  Groups: Group 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of ozanimod vs azathioprine for the treatment of ulcerative colitis (UC) in real-world clinical practice in Japan

ELIGIBILITY:
Inclusion Criteria:

* Participants with Ulcerative Colitis (UC) provided written consent to participate in the study
* Participants who are aged ≥ 18 years at the earlier date of either initiation of treatment with ozanimod or azathioprine or obtaining consent
* Starting dose of oral steroid ≥ 30 mg/day (prednisolone equivalent)
* Administration of ozanimod or azathioprine started after oral steroid administration, and ozanimod or azathioprine administered concomitantly with steroids (excluding patients who started oral steroids and ozanimod or azathioprine on the same day)
* In the ozanimod group, patients with notable clinical symptoms due to the primary disease (rectal bleeding subscore ≥ 1 point or total PRO2 score ≥ 2 points) remained at the start of ozanimod administration
* In the azathioprine group, patients who started azathioprine treatment after February 2019

Exclusion Criteria:

* Participants with symptoms of UC with no change or increase in Patient-Reported Outcome 2 (PRO2) from the time of initiating oral steroid administration after 2 weeks of administration of ≥ 30 mg/day (prednisolone equivalent) of oral steroids
* Participants with complications requiring continued steroid use (excluding topically acting steroids for inhalation or topical application)
* Participants who participated in other clinical studies involving interventions during the observation period
* Participants judged to be inappropriate for enrollment in this study by the investigator at each participating study site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults diagnosed with ulcerative colitis (UC) who initiated ozanimod or azathioprine treatment after starting oral steroids and concomitant-use oral steroids in Japan
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving steroid-free symptomatic remission | Week 12; Weeks 24 and 52

SECONDARY OUTCOMES:
Oral steroid dose prescribed | Week 12; Weeks 24 and 52
Proportion of patients with continuation of ozanimod or azathioprine treatment after oral steroid treatment initiation | Weeks 24 and 52
Steroid-free maintenance period duration | Up to Week 52
Time to achieving steroid-free status | Up to Week 52
Incidence of adverse events (AEs) and treatment-related adverse events (TRAEs) | Up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Sapporo Medical university school of Medicine, Hokkaidō, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts